CLINICAL TRIAL: NCT03022500
Title: Phase II Study of Durvalumab + Tremelimumab in Pulmonary Sarcomatoid Carcinoma
Brief Title: Pulmonary sarcomatoid_MEDI4736+Treme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Bhumsuk Keam, Clinical Assistant Professo, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSC
Record Dates: First submitted 2017-01-13; First posted 2017-01-16 (Estimated); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Durvalumab + Tremelimumab Combination Treatment, Pulmonary Sarcomatoid Carcinoma, NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- durvalumab + tremelimumab (Experimental): Durvalumab: 1.5g Q4W plusTremelimumab: 75mg Q4W up to 4cycle then Durvalumab 750mg Q2W, till PD or unacceptable toxicity.
  Interventions: Drug: durvalumab + tremelimumab

INTERVENTIONS:
Drug: durvalumab + tremelimumab — Durvalumab: 1.5g Q4W plus Tremelimumab: 75mg Q4W up to 4cycle then Durvalumab 750mg Q2W, till PD or unacceptable toxicity.

SUMMARY:
To understand efficacy of Durvalumab(MEDI4736)+ Tremelimumab in Metastatic/relapsed pulmonary sarcomatoid carcinoma

DETAILED DESCRIPTION:
This is a phase II multi-center, open-label study to evaluate efficacy and safety of durvalumab + tremelimumab combination treatment in patients with pulmonary sarcomatoid carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20 years
2. ECOG PS ≤1
3. Patients with histologically confirmed NSCLC with the histology of sarcomatoid carcinoma (WHO criteria for sarcomatoid carcinoma is used; Carcinoma with spindle and/or giant cells, Pleomorphic carcinoma, Spindle cell carcinoma, Giant cell carcinoma, Carcinosarcoma, pulmonary blastoma. If the NSCLC patients showed sarcomatoid carcinoma histology in re-biopsy sample(so called epithelial-mesenchymal transition (EMT) phenomenon),the patients are eligible)
4. Initial metastatic cases or recurrent cases after curative treatment (any chemotherapy line is allowed)
5. A patient with at least one measurable lesion of which the diameter is confirmed to be ≥ 10mm in spiral CT or multi-detector CT (MD CT), or ≥ 20 mm in conventional CT (it should be used by a consistent method during the study period).
6. If patients have brain metastasis with neurological symptom, they should be stabilized neurologically with prior radiotherapy or surgery for the brain metastasis (no neurologic symptom in progress and without further steroid treatment)
7. Adequate hematologic (neutrophil count ≥ 1,500 cells/mm3, platelets ≥ 100,000 cells/mm3), hepatic (transaminase ≤ upper normal limit(UNL)x2.5, bilirubin level ≤ UNLx1.5), and renal (creatinine ≤ UNL) function
8. A patient with the willingness to comply with the study protocol during the study period and capable of complying with it.
9. A patient who signed the informed consent prior to the participation of the study and who understands that he/she has a right to withdrawal from participation in the study at any time without any disadvantages - Absolute neutrophil count 1,500 cells/mm3, platelets 100,000 cells/mm3
10. Expected survival ≥ 3 months
11. Female subjects must either be of non-reproductive potential (ie, post-menopausal by history: ≥60 years old and no menses for ≥1 year without an alternative medical cause; or history of hysterectomy, or history of bilateral tubal ligation, or history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.

Exclusion Criteria:

1. A patient with no measurable disease
2. chronic systemic steroid therapy or on any other form of immunosuppressive medication
3. has received a live-virus vaccination within 30 days of planned treatment start
4. history of diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction, abdominal carcinomatosis which are known risks factors for bowel perforation
5. active symptomatic central nervous system (CNS) metastases and/or carcinomatous meningitis
6. severe hypersensitivity reaction to treatment with another monoclonal antibody (mAb)
7. active autoimmune disease within the past 2 years (NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment -within the past 2 years- are not excluded) or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents
8. prior treatment with any other anti-programmed cell death protein-1 (anti-PD-1), or PD Ligand-1 (PD-L1) or PD Ligand-2 (PD-L2) agent or anti CTLA4 agents (including durvalumab and tremelimumab)
9. active infection requiring therapy
10. history of Human Immunodeficiency Virus (HIV)
11. active Hepatitis B or C (inactive healthy carriers of HBV with appropriate prophylactic antiviral agents are allowed)
12. symptomatic ascites or pleural effusion
13. pneumonitis that has required a course of oral steroids to assist with recovery, or a history of interstitial lung disease
14. pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study
15. History of active tuberculosis
16. History of allogeneic organ transplant. Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab or tremelimumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
17. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) ≤ 21 days prior to the first dose of study drug
18. History of allogeneic organ transplant
19. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
20. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Response rate (RR) | 12 months after the first date of treatment
  According to modified RECIST1.1, The duration from the first date of treatment to the date of death from any cause or follow-up

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 12 months after the first date of treatment
  The percentage of patients who have not experienced disease progression or death from any cause within 12 months from the start of treatment.
Overall Survival (OS) | 12 months after the first date of treatment
  The duration from the first date of treatment to the date of death from any cause or follow-up
Safety | 12 months after the first date of treatment
  The number of patients with treatment-related AE as assessed by NCI CTCAE version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Bhumsuk Kim, Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Department of Internal Medicine, Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
anticipated as research paper